CLINICAL TRIAL: NCT06275854
Title: Young Adult Survivors United Cancer Research Registry
Brief Title: YASU Research Registry: For Young Adults With Cancer
Status: Terminated | Type: Observational
Why Stopped: Sponsoring organization no longer desired to recruit/maintain registry
Sponsor: Young Adult Survivors United (Other)
Collaborators: Staunton Farm Foundation (Unknown); Elsie H. Hillman Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 22265
Record Dates: First submitted 2024-01-22; First posted 2024-02-23 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Leukemia; Sarcoma; Germ Cell Cancer; Lymphoma; Colorectal Cancer; Melanoma; Breast Cancer
Keywords: young adult cancer
MeSH Terms: conditions — Neoplasms; Leukemia; Sarcoma; Neoplasms, Germ Cell and Embryonal; Lymphoma; Colorectal Neoplasms; Melanoma; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational research registry is to learn about health, wellbeing, and needs of survivors of young adult cancer (diagnosed between the ages of 18 and 39). The main question[s] it aims to understand are:

* What are the levels of depression, anxiety, social support, and financial distress
* Determine effectiveness of YASU programming by measuring changes over time

With this registry, the investigators also plan to identify survivors who may be eligible for participation in future research studies pertaining to young adult cancer.

Participants will be asked to complete electronic surveys every 6 to 12 months during participation in the registry.

DETAILED DESCRIPTION:
The study will be conducted online.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer diagnosis received between the ages of 18 and 39.
2. Able to speak and read English

Exclusion Criteria:

1. Inability to provide consent (such as neurological illness or mental incapacity)
2. Has not registered as a member of YASU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any young adult diagnosed with cancer between the ages of 18 and 39 willing to register on the YASU website and consents to participation in the research registry.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Anxiety | enrollment in registry, 6 months later, yearly until death
  General Anxiety Disorder-7 (GAD-7). Scores range from 0-21 with higher scores indicating higher levels of anxiety.
Depressive symptoms | enrollment in registry, 6 months later, yearly until death
  Patient Health Questionnaire- 9 (PHQ-9) Scores range from 0-27, with higher scores indicating more depressive symptoms.
Social Support | enrollment in registry, 6 months later, yearly until death
  MOS Social Support Survey Instrument The survey consists of four separate social support subscales and an overall functional social support index. A higher score for an individual scale or for the overall support index indicates more support.
  MOS Social Support Survey Instrument
  Measure of Social Support Survey Instrument
Financial Toxicity | enrollment in registry, 6 months later, yearly until death
  COST: A FACIT Measure of Financial Toxicity (COST - FACIT (Ver 2)) Scores range from 0-44. The higher the score, the better the Financial Well-Being
Needs Assessment | enrollment in registry
  AYA Psycho-Oncology Screening Tool (AYA-POST) There is no scoring required for this tool.

SECONDARY OUTCOMES:
Name, address, email, phone number | enrollment in registry
  Contact information if willing to be alerted about future research

CONTACTS AND LOCATIONS:
Locations (1):
- Young Adult Survivors United, Wexford, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Starting once enrollment has been open for 6 months.
Access Criteria: In order to be granted access to our dataset, the outside researcher would need to secure IRB approval for their proposed study and then would sign a YASU-provided confidentiality agreement.
  Datasets shared with researchers outside of YASU will not include identifiers.
  Future research collaborators outside of YASU may use the registry to contact participants for other studies and may have access to screen for candidates. Outside researchers who wish to use contacts from the YASU research registry in recruitment for their study will be required to secure IRB approval for their proposed study and to complete the YASU-provided confidentiality agreement prior to any possible participant contact information being shared. Once IRB-approval has been received and the agreement is completed, the PI (and/or YASU executive director) may grant the requestor access to the requested information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT06275854/Prot_SAP_000.pdf